CLINICAL TRIAL: NCT05469763
Title: Effect of Circuit Training on Calcium Level and Physical Fittness in Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shorouk Ahmed Mohamed Wahb, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003729
Record Dates: First submitted 2022-07-03; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circuit training exercise plus calcium tablets group (Experimental): Study Group: they will receive circuit training exercise, 3 sessions per week for 12 weeks, in addition to calcium supplements.
  Interventions: Other: Circuit training
- Calcium tablets group (Other): Control Group: they will receive daily dosage of calcium supplements 1-3 g/ day
  Interventions: Other: Circuit training

INTERVENTIONS:
Other: Circuit training — Mode : any rhythmical and aerobic activity using large muscle groups that can be maintained continuously.
  * Intensity: 60% to 90% of maximum heart rate reserve or 50% to 85% of vO2 max.
  * Duration: 25 to 30 minutes of continuous aerobic activity.
  * Frequency: three to five days per week.

SUMMARY:
This study will be conducted to determine the effect of circuit weight training on calcium level and physical fitness in pregnant

DETAILED DESCRIPTION:
During pregnancy, hem-dilution causes the serum albumin and hemoglobin to decrease. This fall in albumin causes the total serum calcium to fall to levels normally associated with symptomatic hypocalcaemia. The deficiency also occurs due to low dietary intake of calcium .This deficiency has a negative effect on both the mother and the fetus, as high blood pressure , maternal hypocalcemia, abortion, numbness and tingling in the fingers, muscle and leg cramps, poor appetite, heart problems, premature birth, low birth weight, perinatal death, and neonatal tetany .

General physical exercises specially circuit weight training will aids to increase calcium level as it plays a major role in increasing bone density not only through mechanical loading ,but also through blood PH and biomechanical changes in free ionized calcium, which can positively affect bone density . Circuit weight training exercises can improve the health related physical fitness variables namely cardiovascular fitness , muscular strength, muscular endurance, flexibility , balance and speed

Various studies investigated the effect of circuit weight training on bone mineral density and its effect on improving general fitness but there is a gap in the literature of review about its effect on calcium level and physical fitness in gravid women .So, this study will be of valuable benefits for medical service organizations and increase body of knowledge for physical therapists in women's health field.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women suffering from a decrease in blood calcium level, (<500 mg) dietary intake as recorded by food frequency questionnaire.
* They will be selected at second trimester (18th-24thweeks).
* Their age will range from (20 to 35) years old.
* Their BMI will be (35.00 to39.99) Kg/m2 in the second trimester.

Exclusion Criteria:

* Highly risk pregnant women (gestational diabetes &pre-eclampsia).
* Pregnant women with risk for pre-term labor.
* Pregnant women with a history of habitual abortion.
* Pregnant women with thyroid, kidney and liver dysfunction and women with cardiovascular diseases.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Calcium levels | Up to 2 months
  * Total calcium
  * Ionized calcium
  * Free calcium
  will be measured before and after the study program for pregnant women in both groups.

SECONDARY OUTCOMES:
Sit and reach flexibility test | Up to 2 months
  The pregnant woman will perform a short warm up before performing a fitness testing. This test measures the flexibility of the lower back and hamstring muscles. The equipment required will a special testing box and ruler. The procedure of this test involves sitting on the floor with legs stretched out straight ahead. After some practice reaches, the participating woman reaches out and holds that position for one-two seconds while the distance is recorded. Three trials will be given to the participating woman and the highest scores will be recorded.
Modified push up test for upper body endurance | Up to 2 months
  The pregnant woman will perform a short warm up before performing a fitness testing. Push up measure the muscular endurance of the upper body muscles to include the shoulders, chest and back of the upper arms. This fitness area is related to the use of force involving pushing motion. Modified push up will be performed with flexed knee and continued until failure (e.g. inability to continue due to muscle fatigue). Recruits assume a push up position with feet together or up to twelve inches apart. Hands will placed approximately shoulder width apart with fingers facing forward. A partner recruit will be in a position to extend a fist on the floor directly underneath the testing recruit's sternum. A proper push up is when the testing recruit lowers the body and touches the fist with sternum then returns up to the starting position with the elbows in a soft lock. Proper form is closely monitored. Three trails will be given to the participating woman and the highest will be recorded.
Wall squat test for muscular strength | Up to 2 months
  The pregnant woman will perform a short warm -up before performing a fitness testing. This test will be used to test the quadriceps strength. To undertake this test the researcher requires a warm dry location-gym, smooth wall, stopwatch assistant. The Wall Squat test will be conducted as follows, the participating woman will stand comfortable on both feet with back against a smooth wall slide back down the wall, there is to be a 90°angle at the hip and knee, when the participating woman is ready lift one foot 5cm off the ground, the assistant starts the stopwatch as long as possible. The watch is stopped when they put their foot back on the ground; the researcher takes a test and then repeats the test with the other leg. The best time result will be recorded as a score in the second.
Chair stand test for muscular fitness | Up to 2 months
  This test measures leg strength and endurance. The equipment required is a straight back or folding chair without arm rests (seat 17 inches/ 44 cm high). Place the chair against a wall , or otherwise stabilize it for safety. The pregnant woman will sit in the middle of the seat , with her feet shoulder width apart, flat on the floor. The arms will be crossed at the wrists and held close to the chest. From the sitting position , she will stand completely up, then completely back down , and this will be repeated for 30 seconds.
Steady state test for cardiovascular fitness | Up to 2 months
  This test measures how you can maintain your effort for longer periods. This test is sustained for an extended time usually starting at about 10 to 15 minutes at a fixed intensity. In this study we will choose walking form. The pregnant woman will be start with 15 minutes and shoot for a target heart rate of lower than 55% of her maximum heart rate. Gradually she will be increase her steady state training to a 20 minutes cardio routine , eventually going up to 30 minutes.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF